CLINICAL TRIAL: NCT00982579
Title: An Open Randomized Phase I Study Evaluating Safety and Immunogenicity of a Candidate HIV-1 Vaccine, MVA.HIVA, Administered to Healthy Infants Born to HIV-1/2-uninfected Mothers
Brief Title: Safety and Immunogenicity Study of Candidate HIV-1 Vaccine Given to Healthy Infants Born to HIV-1/2-uninfected Mothers
Acronym: PedVacc001
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medical Research Council (Other Government)
Collaborators: European and Developing Countries Clinical Trials Partnership (EDCTP) (Other Government)
Responsible Party: Dr. Tomas Hanke, Medical Research Council, UK
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PV001
Record Dates: First submitted 2009-09-22; First posted 2009-09-23 (Estimated); Last update posted 2012-02-03 (Estimated); Status verified 2009-09

CONDITIONS: HIV-1; HIV Infections
Keywords: HIV preventive vaccine
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vaccinees (Experimental): Vaccinated at 20 weeks of age (n=24)
  Interventions: Biological: MVA.HIVA
- Controls (No Intervention): No experimental vaccine (n=24)

INTERVENTIONS:
Biological: MVA.HIVA — 1 dose of 5 x 10^7 pfu of MVA.HIVA administered intramuscularly
  Arms: Vaccinees

SUMMARY:
Objectives:

Safety and immunogenicity of MVA.HIVA vaccine in 20-week-old healthy Gambian infants born to HIV-1/2-uninfected mothers.

Gross impact of MVA.HIVA on the immunogenicity of EPI vaccines (DTwPHib, HepB, PCV-7 and OPV) when administered at 20 weeks (4 weeks after the last EPI vaccines), who have had BCG vaccine within the first 4 weeks of life.

ELIGIBILITY:
Inclusion Criteria:

* Healthy infants, 19 weeks of age, with weight for age z-scores within 2 standard deviations of normal.
* Have received all standard EPI immunizations according to national immunization programme.
* Written informed consent by parent.
* Mother HIV-1/2-uninfected.

Exclusion Criteria:

* Acute disease at the time of vaccination (acute disease is defined as the presence of a moderate or severe illness with or without fever). All vaccines can be administered to persons with a minor illness such as diarrhoea, mild upper respiratory tract infection with or without low-grade febrile illness, i.e. axillary temperature of <37.5 °C ).
* Axillary temperature of ≥ 37.5 °C at the time of vaccination.
* Any clinically significant abnormal finding on screening from biochemistry or haematology at 19 weeks.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine, e.g. egg products.
* Presence of any underlying disease that compromises the diagnosis and evaluation of response to the vaccine.
* Invasive bacterial infections (pneumonia, meningitis).
* Any other on-going chronic illness requiring hospital specialist supervision.
* Administration of immunoglobulins and/or any blood products within one month preceding the planned administration of the vaccine candidate.
* Any history of anaphylaxis in reaction to vaccination.
* Research physician's assessment of lack of willingness by parents to participate and comply with all requirements of the protocol, or identification of any factor felt to significantly increase the infant's risk of suffering an adverse outcome.
* Likelihood of travel away from the study area.
* Untreated malaria infection.
* Any other clinical evidence of infection.

Max Age: 3 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2009-11; Primary Completion 2011-06 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
For safety and reactogenicity: Actively and passively collected data on adverse events | Up to 16 weeks after vaccination

SECONDARY OUTCOMES:
For immunity to EPI vaccines: Antibody levels to specific vaccines. | 1 week before and 1 week after vaccination
For immunogenicity: Frequency of IFN-γ producing cells determined in ex-vivo (effector) and 10-day cultured (memory) ELISPOT assays after overnight stimulation with pools of HIVA-derived peptides | Up to 16 weeks after vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Tomas Hanke, Study Director — Medical Research Council; Katie Flanagan, Principal Investigator — Medical Research Council, The Gambia; Marie Reilly, Principal Investigator — Karolinska Institutet
Locations (1):
- Medical Research Council Laboratories, The Gambia, Banjul, Fajara, The Gambia

REFERENCES:
- [Derived] Afolabi MO, Ndure J, Drammeh A, Darboe F, Mehedi SR, Rowland-Jones SL, Borthwick N, Black A, Ambler G, John-Stewart GC, Reilly M, Hanke T, Flanagan KL. A phase I randomized clinical trial of candidate human immunodeficiency virus type 1 vaccine MVA.HIVA administered to Gambian infants. PLoS One. 2013 Oct 24;8(10):e78289. doi: 10.1371/journal.pone.0078289. eCollection 2013. PMID 24205185